CLINICAL TRIAL: NCT07163117
Title: The Efficacy of Lumber Stabilization Exercise Versus Back Endurance Exercise on the Range of Motion of the Lumber Spine and Its Stability Among Female University Students
Brief Title: Lumber Stabilization Exercise Versus Back Endurance Exercise Among Female University Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7419
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: stabilization exercises; range of motion; endurance training; lumber spine
MeSH Terms: interventions — Endurance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Lumbar stabilization group) (Experimental): This group will receive lumbar stabilization exercises in addition to home based program two times per week for four consecutive weeks.
  Interventions: Other: lumbar stabilization exercises; Other: Home based program
- Group B (Trunk endurance) (Experimental): This group will receive trunk endurance exercises for back flexors and extensors in addition to home based program two times per week for four consecutive weeks.
  Interventions: Other: endurance training; Other: Home based program
- Group C (control group) (Active Comparator): This group will receive home based program two times per week for four consecutive weeks.
  Interventions: Other: Home based program

INTERVENTIONS:
Other: lumbar stabilization exercises — The participants required to be in a prone position with pillow under abdomen, first raise one leg then the other leg, raise one arm then the other arm, after that raise two legs together, then raise two arms together, raise right arm with left leg then left arm with right leg, then raise both arms and both legs together, every position hold for 20 seconds. Then they required to be in a half kneeling on standing for right leg hold for 20 second and repeat for other leg, do it again but their knees doesn't touch the ground. Finally they required to lie on their backs, and bend their knees at around a 90 degree angle. Place their hands to their sides and their feet flat on the floor at about shoulder width and asked to raise their hips off the floor, hold 20 second.
  Arms: Group A (Lumbar stabilization group)
Other: endurance training — 1. Back extensor endurance training exercise:
     The participants lay prone over the end of a treatment table with the anterior superior iliac spine supported on the bench edge. Their ankles were fixed by the researcher. They maintained the horizontal position for as long as possible, beginning timing when the horizontal unsupported position was achieved and ending when they dropped below the horizontal plane. The duration of holding was measured in seconds.
  2. Back flexor endurance training exercise:
  The participants asked to sit on the table with your arms crossed against their chest and their back against the wedge. Fix them to the table with a belt across the feet. They asked to remove the wedge from their back using the timing device to record how much time is accumulated until the original position can no longer be maintained.
  Arms: Group B (Trunk endurance)
Other: Home based program — General and similar exercises for back muscles introduced for this group. They instructed to do knee to chest stretch, lower back rotational stretch, bridge exercise. The required measure data were obtained from the selected cases in this group before and after the end of rehabilitation program.

SUMMARY:
Low Back Pain (LBP) as estimates show that up to 84% of adults will experience LBP at some point in their lifetime, ranking it as a leading cause of disability globally. If the pain lasts more than 12 weeks and remains difficult to manage effectively, it can be called Chronic low back pain (CLBP). Physical therapy interventions play an important role in the non-pharmacological management of CLBP including lumbar stabilization exercises (LSEs) and back extension/endurance exercises which are commonly prescribed modalities that may help in improving the spinal function, reducing pain and improving the quality of life in general.

DETAILED DESCRIPTION:
LSEs can be considered as an isometric contraction that might be used to strengthen the deep core muscles surrounding the lumbar spine. Studies showed that although most conventional therapies can improve lumbar stability and reduce the severity of CLBP, LSEs are the most effective technique. However, both back extension and endurance exercises can play a significant role in strengthening the superficial back muscles particularly in the lower back region via dynamic movements.

ELIGIBILITY:
Inclusion Criteria:

* BMI ranged from 28 to 29 kg/ cm2.
* clinically diagnosed by an orthopedic consultant as having a history of mechanical low back pain for at least three months.

Exclusion Criteria:

* Previous trauma.
* Previous surgery.
* Any musculoskeletal disorder
* Any neurological disorder (disc prolapse, or spondylosis)

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Spinal range of motion (ROM) | 4 weeks
  Two inclinometers will be used. One placed at T12-L1 (thoracic 12- lumbar 1) and another placed at L5-S1 (lumbar 5-sacrum 1), respectively.

SECONDARY OUTCOMES:
Trunk Endurance | 4 weeks
  Endurance test will be performed in flexion and extension using stop watch to record how long the patient can maintain these two positions.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 6 months after publication